CLINICAL TRIAL: NCT04857684
Title: A Pilot Study of Neoadjuvant Stereotactic Beam Radiation Therapy Followed by Atezolizumab and Bevacizumab in Resectable Hepatocellular Carcinoma
Brief Title: SBRT + Atezolizumab + Bevacizumab in Resectable HCC
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Jennifer Wo, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-570
Record Dates: First submitted 2021-04-16; First posted 2021-04-23 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma; Resectable Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Resectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stereotactic beam radiation therapy (SBRT) +Atezolizumab + Bevacizumab (Experimental): Participants will:
  * undergo a pre-treatment biopsy with fiducial marker placement
  * receive Stereotactic beam radiation therapy (SBRT) on three treatment days which will be arranged on an every-other-day basis
  * receive two 3-week (21 days) cycles of atezolizumab plus bevacizumab
    * receive Atezolizumab on day 1 for 2 study cycles.
    * receive Bevacizumab 1x weekly for 2 study cycles
  * Surgery after SBRT and the two cycles of atezolizumab and bevacizumab, unless participants are otherwise informed by their doctor. The planned surgery will take place 6-8 weeks after the last infusions of atezolizumab and bevacizumab.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Radiation: Stereotactic Beam Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: Atezolizumab — Intravenous Infusion
  Other Names: Tecentriq
Drug: Bevacizumab — Intravenous Infusion
  Other Names: Avastin
Radiation: Stereotactic Beam Radiation Therapy (SBRT) — External beam radiation
  Other Names: Radiation Therapy

SUMMARY:
This study is evaluating the safety and tolerability of neoadjuvant stereotactic body radiation therapy (SBRT) with atezolizumab and bevacizumab for treating resectable hepatocellular carcinoma.

This study involves the following study interventions:

* Atezolizumab
* Bevacizumab
* Stereotactic Beam Radiation Therapy (SBRT)
* Surgery

DETAILED DESCRIPTION:
This is a single-center, open-label, single-arm pilot study designed to evaluate the safety and tolerability of neoadjuvant radiation therapy plus atezolizumab and bevacizumab in patients with treatment-naïve resectable hepatocellular carcinoma.

This research study is a Pilot Study, which is the first-time investigators are examining this intervention of neoadjuvant radiation therapy plus atezolizumab and bevacizumab.

The U.S. Food and Drug Administration (FDA) has not approved atezolizumab, bevacizumab, stereotactic body radiation therapy (SBRT) for resectable hepatocellular carcinoma but they have been approved for other uses. Surgery is an accepted and standard treatment option for resectable hepatocellular carcinoma

The study interventions (atezolizumab bevacizumab, and SBRT) are thought to increase the immune system's (the system in the body that fights against disease) response to cancer cells. These interventions may increase the immune system's response by helping the T cells (an immune cell that identifies and attacks infected cells) recognize and find cancer cells in the body. By increasing the system's response, it is believed the chances of recurrence of resectable hepatocellular carcinoma will be less than when only standard of care surgery is used.

The research study procedures include screening for eligibility and study treatment, including evaluations and follow up visits.

Participants will receive study treatment for as long as they and their doctor believe they are benefitting from the study interventions and will be followed for 5 years or until participants withdraw their consent to be contacted.

It is expected that about 20 people will take part in this research study

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of hepatocellular carcinoma that is localized to the liver, has no radiographic evidence of macrovascular invasion, and is deemed surgically resectable. The diagnosis may be obtained radiographically (i.e. having a LiRADS or OPTN category 5 liver lesion) or by histologic diagnosis from a core biopsy or cytology specimen. Radiographic evaluation should occur within approximately 30 days prior to enrollment.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam. See Section 12 (Measurement of Effect) for the evaluation of measurable disease.
* Participants must have Child-Pugh A liver function (see Appendix A).
* No prior therapy directed against the index hepatocellular carcinoma lesion is allowed
* Age ≥18 years at the time of signing the informed consent document.
* ECOG performance status ≤ 1 (Karnofsky ≥60%, see Appendix B).
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ 2 × institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
  * creatinine ≤ 1.5 × institutional ULN OR
  * estimated glomerular filtration rate (GFR) ≥50 mL/min/1.73 m2 (according to the Cockcroft-Gault formula)
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Documented virology status of hepatitis, as confirmed by screening tests for HBV and HCV

  * For patients with active HBV: HBV DNA <500 IU/mL during screening, initiation of anti-HBV treatment at least 14 days prior to randomization and willingness to continue anti-HBV treatment during the study (per local standard of care; e.g., entecavir)
  * Patients with HCV, either with resolved infection (as evidenced by detectable antibody and negative viral load) or chronic infection (as evidenced by detectable HCV RNA), are eligible.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* The effects of the combination of radiation and atezolizumab plus bevacizumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to either abstain from sexual intercourse or use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of atezolizumab and bevacizumab administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed/biphenotypic cholangiocarcinoma-HCC.
* Radiographic evidence of metastasis to lymph nodes or other extra-hepatic sites.
* History of hepatic encephalopathy, moderate or severe ascites.
* Coinfection with HBV and HCV. Patients with a history of HCV infection but who are negative for HCV RNA by PCR will be considered non-infected with HCV.
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or that are at high risk for bleeding Patients must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed and treated per local standard of care prior to enrollment. Patients who have undergone an EGD within 6 months of prior to initiation of study treatment do not need to repeat the procedure.
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment
* Inadequately controlled hypertension, defined as systolic blood pressure (BP) <150 mmHg and/or diastolic BP < 100 mmHg (average of at least three readings at two or more sessions). Anti-hypertensive therapy to achieve these parameters is allowed.
* History of hypertensive crisis or hypertensive encephalopathy.
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to initiation of study treatment
* History of hemoptysis (> 2.5 mL of bright red blood per episode) within 1 month prior to initiation of study treatment
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Current or recent (< 10 days prior to initiation of study treatment) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose. Prophylactic anticoagulation for the patency of venous access devices allowed, provided the activity of the agent results in an INR < 1.5 x ULN and aPPT is within normal limits within 14 days prior to initiation of study treatment. For prophylactic use of anticoagulants or thrombolytic therapies, the approved dose as described on the local label may be used.
* Current or recent (< 10 days prior to initiation of study treatment) use of aspirin (> 325 mg/day) or treatment with clopidogrel, dipyramidole, ticlopidine, or cilostazol.
* Participants who are receiving any other investigational agents.
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 3 days prior to initiation of study systemic therapy.
* History of abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months prior to initiation of study treatment.
* History of intestinal obstruction and/orclinical signs or symptoms of GI obstruction, including subocclusive or occlusive syndrome related to the underlying disease, or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding prior to initiation of study systemic therapy. Patients with signs or symptoms of subocclusive or occlusive syndrome or with intestinal obstruction at the time of initial diagnosis may be enrolled if they had received definitive (surgical) treatment for symptom resolution.
* Evidence of abdominal free air that is not explained by paracentesis or other recent surgical or interventional procedure.
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture.
* Grade 2 proteinuria, as demonstrated by 2+ protein on dipstick urinalysis and 1.0 g of protein on a 24-hour urine collection. All patients with 2+ protein on dipstick urinalysis at screening must undergo a 24-hour urine collection for protein. Patients with 2+ protein on dipstick urinalysis are eligible for the study.
* Patients with vascular invasion of the portal veins may NOT be enrolled, with the exceptions of patients with vp1 tumor thrombus (involvement distal to the second-order branches of the portal vein).
* History of intra-abdominal inflammatory process within 6 months prior to initiation of study treatment, including but not limited to: peptic ulcer disease, diverticulitis, or colitis.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to initiation of study treatment; or abdominal surgery, abdominal interventions, or significant abdominal traumatic injury within 60 days prior to initiation of study treatment.
* Chronic daily treatment with a nonsteroidal anti-inflammatory drug (NSAID). The occasional use of NSAIDs for the symptomatic relief of medical conditions such as headache or fever is allowed.
* Active or history of autoimmune disease or immune deficiency, inclusing but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel diseae, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis. Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for this study. Patients with type I diabetes mellitus are eligible for this study. Patients with eczema, psoriasis,lichen simplex chronicus, or vitiligo with dermatologic manifestations (e.g. patients with psoriatic arthritis are exluded) are eligible for the study provided that all of the following conditions are met:

  * Rash must cover <10% of body surface area
  * Disease is well-controlled at baseline and requires only low-potency topical corticosteroids.
  * No occurrence or acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screen chest computed tomography (CT) scan.
* Active tuberculosis (TB) as documented by a positive purified protein derivative (PPD) skin test or TB blood test and confirmed by a positive chest radiograph within 3 months prior to initiation of study treatment. Patients with a positive PPD skin test or TB blood test followed by a negative chest radiograph may be eligible for the study.
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study.
* History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
* Prior allogeneic stem cell or solid organ transplantation or on the wait list for liver transplantation.
* Pregnancy or breastfeeding, or intending to become pregnant during the study. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment. The rationale for this exclusion is the unknown toxicities of immune checkpoint inhibitors on developing fetuses and the known placental risk conferred by treatment with vascular endothelial growth factor inhibitors (such as bevacizumab).
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
* Known hypersensitivity to Chinese hamster ovary cell products or recombinant human antibodies.
* Known allergy or hypersensitivity to any of the study drugs or any of their excipients.
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment.
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Medical Monitor confirmation has been obtained.
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* Since this study aims to enroll only resectable (with curative intent) hepatocellular carcinoma subjects, patients with brain (or other sites of distant) metastases are excluded.
* Participants with uncontrolled intercurrent illness.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2027-04-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with grade 3-4 treatment-related adverse events as assessed by CTCAE v5.0 | From enrollment to end of treatment, up to 6 months
  Assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Objective response rate (ORR) | From enrollment to end of treatment, up to 3 months
  Assessed by RECIST 1.1
Proportion of patients who proceed to surgery after neoadjuvant treatment. | From enrollment to end of treatment, up to 3 months
  Estimated with 95% confidence intervals based on the exact binomial distribution.
Proportion of patients who undergo a microscopic margin-negative (R0) resection | From enrollment to end of treatment, up to 3 months
  Estimated with 95% confidence intervals based on the exact binomial distribution.
Complete response (CR) | From enrollment to end of treatment, up to 3 months
  Assessed by RECIST 1.1
Overall survival (OS) | From enrollment to end of treatment, up to 2 years
  Estimated by the Kaplan-Meier method
Recurrence-free survival (RFS) after resection | From enrollment to end of treatment, up to 2 years
  Estimated by the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Y Wo, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation